CLINICAL TRIAL: NCT02129842
Title: A Prospective, Non-randomized, Double Blind Multicenter Study to Assess Endothelial Function Using Endo-PAT2000 and Its Correlation to Clinical Outcome Following Ablation in Patients With Atrial Fibrillation
Brief Title: Is Endothelial Function a Predictor of Successful Ablation Therapy Provided to Patients With Atrial Fibrillation?
Status: Completed | Type: Observational
Sponsor: Itamar-Medical, Israel (Industry)
Responsible Party: Sponsor
Other Study IDs: Endo-AFib-001
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2017-03-09 (Actual); Status verified 2014-12

CONDITIONS: Atrial Fibrillation
Keywords: AFib; AF; ablation; EndoPAT; Endothelial dysfunction; PAT
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Atrial Fibrillation

SUMMARY:
The purpose of this study is to assess whether normal endothelial function in patients with Atrial Fibrillation undergoing ablation procedure increases the chances of a favorable clinical outcome and maintaining sinus rhythm following ablation

DETAILED DESCRIPTION:
In the recent years, increasing evidence is linking inflammation to AFib. In addition, it has been shown that ablation improves endothelial function, suggesting that AFib might be associated with the etiology of endothelial dysfunction.

The objective of this study is to assess endothelial function using Endo-PAT2000 and its correlation to clinical outcome following ablation of patients with Atrial Fibrillation (AFib).

ELIGIBILITY:
Inclusion Criteria:

* All patients with AF considered eligible for ablation treatment may be included in this study (following unsuccessful attempts with AAD).
* Patients on optimal anticoagulation therapy
* The minimum AF documentation required as defined by the Heart Rhythm Society

Exclusion Criteria:

* Patients age below 18 years
* Cases with extremely abnormal anatomy (i.e., inverted heart)
* Moderate or severe mitral valve disease or mitral prosthetic valve
* Ejection fraction less than 30%
* Left atrial anteroposterior diameter more than 50 mm evaluated by echo or CT data (up to 6 months old)..
* Previous atrial fibrillation ablation occurred less than 6 months prior
* Left atrium thrombus
* Acute infective disease or sepsis in the last 3 months
* Acute myocardial infarction in last 3 months
* Reduced expectancy of life (less than 12 months)
* Patient participating in another clinical study that investigates a drug or device unless prior approval is given by the sponsor
* Psychologically unstable patient or denies to give informed consent
* Deformities of the digits of the upper extremities, which preclude adequate signal acquisition
* Patients under the effect of short-acting Nitroglycerin (3 hours washout period)
* Patient suffering from a medical condition prohibiting blood flow occlusion in both arms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AFib patients eligible for ablation treatment
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Freedom from AF/AFL/AT off antiarrhythmic drugs therapy | 12 months

SECONDARY OUTCOMES:
Acute procedural success: Pulmonary veins isolation | 12 months
75% reduction in the number/duration of AFib episodes | 12 months

CONTACTS AND LOCATIONS:
Locations (6):
- United States (3):
  - New York University School of Medicine, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
- University Heart Center Hamburg, Hamburg, Germany
- Sheba Medical Center, Ramat Gan, Israel
- Royal Brompton & Harefield NHS Foundation Trust, London, United Kingdom

REFERENCES:
- [Background] Calkins H, Kuck KH, Cappato R, Brugada J, Camm AJ, Chen SA, Crijns HJ, Damiano RJ Jr, Davies DW, DiMarco J, Edgerton J, Ellenbogen K, Ezekowitz MD, Haines DE, Haissaguerre M, Hindricks G, Iesaka Y, Jackman W, Jalife J, Jais P, Kalman J, Keane D, Kim YH, Kirchhof P, Klein G, Kottkamp H, Kumagai K, Lindsay BD, Mansour M, Marchlinski FE, McCarthy PM, Mont JL, Morady F, Nademanee K, Nakagawa H, Natale A, Nattel S, Packer DL, Pappone C, Prystowsky E, Raviele A, Reddy V, Ruskin JN, Shemin RJ, Tsao HM, Wilber D. 2012 HRS/EHRA/ECAS Expert Consensus Statement on Catheter and Surgical Ablation of Atrial Fibrillation: recommendations for patient selection, procedural techniques, patient management and follow-up, definitions, endpoints, and research trial design. Europace. 2012 Apr;14(4):528-606. doi: 10.1093/europace/eus027. Epub 2012 Mar 1. No abstract available. PMID 22389422
- [Background] Narayan SM, Krummen DE, Clopton P, Shivkumar K, Miller JM. Direct or coincidental elimination of stable rotors or focal sources may explain successful atrial fibrillation ablation: on-treatment analysis of the CONFIRM trial (Conventional ablation for AF with or without focal impulse and rotor modulation). J Am Coll Cardiol. 2013 Jul 9;62(2):138-147. doi: 10.1016/j.jacc.2013.03.021. Epub 2013 Apr 3. PMID 23563126
- [Background] Pokushalov E, Romanov A, Artyomenko S, Turov A, Shugayev P, Shirokova N, Katritsis DG. Ganglionated plexi ablation for longstanding persistent atrial fibrillation. Europace. 2010 Mar;12(3):342-6. doi: 10.1093/europace/euq014. PMID 20173210
- [Background] Boos CJ, Anderson RA, Lip GY. Is atrial fibrillation an inflammatory disorder? Eur Heart J. 2006 Jan;27(2):136-49. doi: 10.1093/eurheartj/ehi645. Epub 2005 Nov 8. PMID 16278230
- [Background] Yoshino S, Yoshikawa A, Hamasaki S, Ishida S, Oketani N, Saihara K, Okui H, Kuwahata S, Fujita S, Ichiki H, Ueya N, Iriki Y, Maenosono R, Miyata M, Tei C. Atrial fibrillation-induced endothelial dysfunction improves after restoration of sinus rhythm. Int J Cardiol. 2013 Sep 30;168(2):1280-5. doi: 10.1016/j.ijcard.2012.12.006. Epub 2012 Dec 24. PMID 23269316